CLINICAL TRIAL: NCT02554188
Title: Effect of Fasting-mimicking Diet on Immunosenescence and Vaccination in Older Adults: A Randomized Clinical Trial
Brief Title: Fasting-mimicking Diet and Immunosenescence
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: USC has an ICOI because the university owns the patent of the interventional dietary supplement.
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Sebastian Brandhorst, Assistant Research Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: HS-16-00467
Record Dates: First submitted 2015-09-15; First posted 2015-09-18 (Estimated); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Immunosenescence
Keywords: Dietary Intervention; Fasting-mimicking; Influenza Vaccines
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines; Vaccines; Diet

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): Participants will receive Seasonal influenza (flu) vaccine.
  Interventions: Biological: Seasonal influenza (flu) vaccine
- Diet (Experimental): Participants will consume 2 cycles of a 5-day low calorie fasting-mimicking diet with approximately 3 weeks of gap period prior to receiving standard Seasonal influenza (flu) vaccine.
  Interventions: Biological: Seasonal influenza (flu) vaccine; Other: Diet

INTERVENTIONS:
Biological: Seasonal influenza (flu) vaccine — Seasonal influenza (flu) vaccine
  * Fluzone Quadrivalent Vaccine (Sanofi Pasteur), for participants ages 50 - 64 years old
  * Fluzone High-Dose (Sanofi Pasteur), for participants ages 65 years and older
  Other Names: Flu shot
Other: Diet — A 5-day low calorie fasting-mimicking diet
  Arms: Diet

SUMMARY:
The objective of this study is to test a Fasting-Mimicking Diet (FMD) for its efficacy on improving immune response to flu vaccination in an older adult population (50-75 years of age).

DETAILED DESCRIPTION:
This is a randomized clinical trial to test the safety and efficacy of the fasting-mimicking diet (FMD) in an elderly population (50-75 years of age) receiving their annual influenza vaccination. The study will include two arms: Control (normal diet) and FMD (2 cycles of 5-day fasting-mimicking diet within two months). Participants both arms will receive the standard influenza vaccine.The primary endpoint is anti-influenza antibody titers measured 4 weeks after flu vaccination. Secondary endpoints include: (1) body composition changes, measured as BMI, waist to hip ratio; (2) physiological changes, measured as blood chemistry and motor performance; (3) health outcomes, measured by SF-36 Health survey, dry eye surveys and flu incidents within 12 months of vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Ability and willingness to provide written informed consent;
* Ability and willingness to undergo 2 cycles of a 5-day dietary regimen;
* Ability and willingness to provide blood samples via venipuncture;
* Seeking to get a seasonal influenza vaccine.

Exclusion Criteria:

Concomitant medications

* Received flu (influenza) shot for the flu season;
* Receiving immunosuppressive therapy (i.e., oral prednisone in doses > 10 mg daily);
* On immunosuppressive drugs for cancer or rheumatologic therapy;
* Receiving insulin or octreotide;
* On hypertension medication. The subject must obtain the treating doctor's approval prior to beginning the study.

Safety-based exclusions:

* Hemoglobin < 9.0 g/dL;
* White blood cell count < 3,500/mm^3;
* Neutrophil count < 2,000/mm^3,
* Platelet count < 125,000/mm^3;
* Medical conditions that are incompatible with the dietary intervention ;
* Medical conditions that are incompatible with the flu vaccination;
* Pregnant or nursing female;
* Alcohol dependency;

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Anti-Influenza Serum antibody titers 4 weeks after flu vaccination | 3 months
  * The ratio of post vaccine to pre vaccine titers will be calculated
  * A positive titer is defined as 1:40 or greater.

SECONDARY OUTCOMES:
Body composition changes | 3 months
  Body composition changes, measured as BMI, waist to hip ratio
Physiological changes | 3-6 months
  Physiological changes measured as blood chemistry and motor performance
Health outcomes | 3-12 months
  Health outcomes measured by SF-36 Health survey.
Flu incidence and severity questionnaire | up to 1 years
  Self-reporting of flu incidence; Self-reporting of flu symptom severity on a 0-5 scale.
Dry eye surveys | up to 1 years
  Dry eye condition measured by the Ocular Surface Disease Index (OSDI) questionnaire and the Dry Dye Severity Questionnaire (DESQ).

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Zelinski, PhD, Principal Investigator — University of Southern California

IPD SHARING:
Plan to Share IPD: No